CLINICAL TRIAL: NCT07214207
Title: Orexin Receptor Antagonism for the Treatment of Alcohol Use Disorder and Stress-Related Drinking
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Stephanie M Gorka, PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20250713; R01AA032711 (NIH)
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: suvorexant; alcohol use disorder; electromyography
MeSH Terms: conditions — Alcoholism | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): Individuals will take a placebo pill daily for 8-weeks.
  Interventions: Other: Placebo
- Suvorexant (Experimental): Individuals will take 10mg of suvorexant (Merck & Co Inc.) daily for 8-weeks.
  Interventions: Drug: Suvorexant 10 mg

INTERVENTIONS:
Drug: Suvorexant 10 mg — This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment, mid-treatment, and post-treatment lab visits. Suvorexant (SUV) will be placed in opaque capsules with dextrose filler. Following the pre-treatment visit, participants will receive a labeled blister pack with 28 pills and be instructed to take one pill orally about 30 minutes prior to sleep time each night for 4 weeks. Participants will be provided education about common side effects. At the end of the 4-weeks, participants will return to the lab to complete a mid-treatment lab visit, receive a second labeled blister pack, and will be instructed to continue taking one pill orally about 30 minutes prior to sleep time each night for 4-weeks. Participants will return to complete a post-treatment lab visit. Participants will complete daily surveys to monitor side effects throughout the 8-week medication trial.
  Other Names: Belsomra
  Arms: Suvorexant
Other: Placebo — This study is a double-blind study. Participants will complete an initial screening visit and pre-treatment, mid-treatment, and post-treatment lab visits. The placebo pill will be identical in appearance to suvorexant but will contain only dextrose. Following the pre-treatment visit, participants will receive a labeled blister pack with 28 pills and be instructed to take one pill orally about 30 minutes prior to sleep time each night for 4-weeks. Participants will be provided education about common side effects. At the end of the 4-weeks, participants will return to the lab to complete a mid-treatment lab visit, receive a second labeled blister pack, and will be instructed to continue taking one pill orally about 30 minutes prior to sleep time each night for 4-weeks. Participants will return to complete a post-treatment lab visit. Participants will complete daily surveys to monitor side effects throughout the 8-week medication trial.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if, how, and for whom suvorexant (SUV) works to treat alcohol use disorder (AUD). The main questions it aims to answer are:

* Is SUV effective for AUD?
* Does SUV dampen stress reactivity?
* Can the researchers develop a biomarker for SUV treatment response?

Researchers will compare SUV to a placebo (a look-alike substance that contains no drug) to see if drug SUV works to treat AUD.

Participants will:

* Take 10mg capsules of SUV or a placebo orally each night before bedtime for 8-weeks.
* Visit the laboratory before (baseline), 4-weeks (mid-point), and 8-weeks (end-point) after taking SUV or placebo that include the psychophysiological stress paradigm (electromyography; EMG).
* Complete daily reports of medication adherence, side-effects, sleep, alcohol use, and mood will be collected via smartphones during the 8-week medication trial.

ELIGIBILITY:
Inclusion Criteria:

* Generally medically and neurologically healthy;
* Age 18 to 65 at the time of consent;
* Willing and able to give informed consent;
* Current DSM-5 diagnosis of moderate to severe alcohol use disorder;
* Engages in heavy alcohol use defined as drinking ≥14 standard drinks per week if male, and ≥7 standard drinks per week if female;
* Self-reported treatment-seeking for alcohol use disorder

Exclusion Criteria:

* Clinically significant medical or neurologic condition or neurocognitive dysfunction that would affect function, and/or task performance, and/or interfere with the study protocol, and/or be contraindicated for suvorexant including sleep disorders (e.g., narcolepsy; severe obstructive sleep apnea), hepatic impairment, compromised respiratory function, renal impairment, and endocrine disorders;
* Lifetime DSM-5 diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder;
* Current substance use disorder (SUD) other than alcohol or mild cannabis use disorder;
* Currently pregnant (positive pregnancy test), lactating, or not agreeing to use birth control methods during the duration of the trial (women);
* Any use of medications for alcohol use disorder or any psychotropic medications (e.g., psychostimulants and benzodiazepines, some antidepressants);
* Current antihistamines use or medication use that may increase risk including, prescribed, over-the-counter, and herbal preparations, as determined by the study physician;
* Current use of strong or moderate inhibitors of CYP3A liver enzymes;
* Current use of strong CYP3A inducers;
* Current use of digoxin;
* Liver function tests more than 3 times the upper limit of normal or elevated bilirubin;
* Engages in night shift work;
* Smoke 10 or more cigarettes (or electronic equivalent) per day and are thus susceptible to acute nicotine withdrawal during lab visits;
* Obesity as defined by a body-mass index (BMI) equal or greater than 30, as calculated from weight and height self-report;
* Clinically significant alcohol withdrawal symptoms the day of the lab sessions, defined as a score >10 on the Clinical Institute Withdrawal Assessment of Alcohol Scale Revised (CIWA-Ar);
* Unwilling/unable to sign the informed consent document;
* Under 18 years old or over 65 years old at the time of enrollment;
* Have attempted suicide in the past 3 years and/or have current suicidal ideation determined as greater than moderate via the Columbia Suicide Severity Rating Scale (C-SSRS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of Heavy Drinking Days | 8-week treatment period
  Self-reported heavy drinking days defined as 5+ drinks for men and 4+ for women. Reported outcome measured as proportion of heavy drinking days.
Startle eyeblink potentiation | Baseline; 4-weeks; 8-weeks
  Startle eyeblink potentiation will be collected during the NPU threat task that is administered at all three lab sessions. Startle is a cross-species index of aversive reactivity.
Alcohol Craving Via Ecological Momentary Assessment (EMA) | 8-week treatment period
  Participants will rate the intensity of their alcohol cravings using a Likert scale of 1 (lowest craving) -7 (highest craving).

SECONDARY OUTCOMES:
Drinks Per Day | 8-week treatment period
  Self-reported total number of alcoholic drinks per day of the trial.
Proportion of Days Abstinent | 8-week treatment period
  Self-reported proportion of days that individuals were abstinent from alcohol use.
Transdermal Alcohol Concentration (TAC) | 8-week treatment period
  Participants' TAC will provide an objective estimate of alcohol consumption each day.
Phosphatidylethanol (PEth) levels | 4-weeks; 8-weeks
  PEth will be measured from plasma samples at the mid-point and end-point. PEth is an objective biomarker of recent alcohol consumption.
Subjective Stress Levels via Ecological Momentary Assessment | 8-week treatment period
  Participants will rate their subjective stress levels using a Likert scale of 1 (least stress) - 5 (most stress).

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this project will be submitted to the NIAAA Data Archive (NDA) at the subject level along with appropriate supporting documentation to enable efficient use of the data by the research community. The investigators will follow instructions as discussed in the NIAAA Data Archive Data Sharing Terms and Conditions.
Time Frame: The data will be submitted to the NIAAA Data Archive biannually per NIAAA requirements throughout the duration of the study.
URL: https://nda.nih.gov/